CLINICAL TRIAL: NCT03130777
Title: Multicenter Study of Congenital Pulmonic Valve Dysfunction Studying the SAPIEN 3 THV With the Alterra Adaptive Prestent
Brief Title: ALTERRA: SAPIEN 3 THV With the Alterra Adaptive Prestent
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-04
Record Dates: First submitted 2017-04-24; First posted 2017-04-26 (Actual); Results first posted 2023-08-08 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Pulmonary Disease; Transcatheter Pulmonary Valve Replacement (TPVR); Tetralogy of Fallot; Congenital Heart Disease; Pulmonary Regurgitation
MeSH Terms: conditions — Lung Diseases; Tetralogy of Fallot; Heart Defects, Congenital; Pulmonary Valve Insufficiency

STUDY DESIGN:
Intervention Model Description: Single arm, prospective, multi-center study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- TPVR - Main Cohort (Experimental): Implantation of Edwards Alterra Adaptive Prestent and Edwards SAPIEN 3 THV using Commander Delivery System.
  Interventions: Device: Edwards Alterra Adaptive Prestent with SAPIEN 3 THV
- TPVR - PDS Registry (Experimental): Implantation of Edwards Alterra Adaptive Prestent and Edwards SAPIEN 3 THV using Pulmonic Delivery System (PDS).
  Interventions: Device: Edwards Alterra Adaptive Prestent with SAPIEN 3 THV

INTERVENTIONS:
Device: Edwards Alterra Adaptive Prestent with SAPIEN 3 THV — The Edwards Alterra Adaptive Prestent is designed to reduce the diameter of large irregular RVOTs and provide a circular, semi-rigid landing zone to place an Edwards SAPIEN 3 THV.

SUMMARY:
To demonstrate the safety and effectiveness of the Edwards Alterra Adaptive Prestent in conjunction with the Edwards SAPIEN 3 Transcatheter Heart Valve (THV) System in subjects with a dysfunctional right ventricular outflow tract/pulmonary valve (RVOT/PV) who are indicated for treatment of pulmonary regurgitation (PR).

Following completion of enrollment, subjects will be eligible for enrollment in the continued access phase of the trial.

ELIGIBILITY:
Inclusion Criteria:

1. The candidate/candidate's legally authorized representative has been informed of the nature of the study, agrees to its provisions and has provided written informed consent.
2. Weight is ≥ 20 kg (44 lbs).
3. RVOT/PV with moderate or greater PR by TTE.
4. RVOT/PV proximal and distal landing zone diameter ≥ 27 mm and ≤ 38 mm, and minimum of 35 mm from contractile tissue to lowest pulmonary artery takeoff.

Exclusion Criteria:

1. Active infection requiring current antibiotic therapy (if temporary illness, patient may be a candidate 2 weeks after discontinuation of antibiotics).
2. History of or active endocarditis (active treatment with antibiotics) within the past 180 days.
3. Leukopenia (WBC < 2000 cells/μL), anemia (Hgb < 7 g/dL), thrombocytopenia (platelets < 50,000 cells/μL) or any known blood clotting disorder.
4. Inappropriate anatomy for introduction and delivery of the Alterra Adaptive Prestent or the SAPIEN 3 THV.
5. Need for concomitant atrial septal defect or ventricular septal defect closure or other concomitant interventional procedures other than pulmonary artery or branch pulmonary artery stenting or angioplasty
6. Interventional/surgical procedures within 30 days prior to the Alterra or valve implant procedure
7. Any planned surgical, percutaneous coronary or peripheral procedure to be performed within the 30 day follow-up from the Alterra or valve implant procedure
8. History of or current intravenous drug use
9. Major or progressive non-cardiac disease resulting in a life expectancy of less than one year
10. Known hypersensitivity to aspirin or heparin and cannot be treated with other antiplatelet and/or antithrombotic medications
11. Known hypersensitivity to nitinol, cobalt-chromium, nickel or contrast media that cannot be adequately pre-medicated
12. Currently participating in an investigational drug or another device study [Note: Trials requiring extended follow up for products that were investigational, but have since become commercially available, are not considered investigational devices.]
13. Positive urine or serum pregnancy test in female patients of child-bearing potential
14. Renal insufficiency (creatinine > 3.0 mg/dL) and/or renal replacement therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2017-08-22 (Actual); Primary Completion 2022-07-14 (Actual); Study Completion 2032-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Evan Zahn, MD, FACC, FSCAI, Principal Investigator — Cedars-Sinai Heart Institute
Locations (14):
- United States (14):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California, Los Angeles, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Emory University/ Children's Healthcare of Atlanta (CHOA), Atlanta, Georgia
  - St. Louis Children's Hospital, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Health Dallas, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas
  - University of Virgina, Charlottesville, Virginia
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Torres AJ, Dimas VV, Shahanavaz S, Balzer D, Morgan G, Lim DS, Armstrong AK, Berman D, Babaliaros V, Kim D, Gillespie MJ, Sommer R, Aboulhosn J, Jones TK, Mahadevan VS, Stapleton G, Ma Y, Shirali G, Parthiban A, Blanke P, Leipsic J, Zahn E. Transcatheter Pulmonary Valve Implantation With the Alterra Adaptive Prestent and SAPIEN 3 Transcatheter Heart Valve: 3-Year Pooled Outcomes of the ALTERRA Trials. Circ Cardiovasc Interv. 2026 Feb 9:e015873. doi: 10.1161/CIRCINTERVENTIONS.125.015873. Online ahead of print. PMID 41657206

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TPVR - Main Cohort | TPVR - PDS Registry
Started | 61 | 25
Completed | 60 | 24
Not Completed | 1 | 1
Not completed — Death | 0 | 1
Not completed — Did not meet eligibility criteria | 1 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Groups:
- Total: Total of all reporting groups
Arm/Group | TPVR - Main Cohort | TPVR - PDS Registry | Total
Number analyzed (Participants) | 61 | 25 | 86
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.5 (16.44) | 29.1 (17.23) | 29.4 (16.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 11 | 38
  Male | 34 | 14 | 48
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Hispanic or Latino | 3 | 2 | 5
  Race: Asian | 5 | 3 | 8
  Race: Black or African American | 7 | 4 | 11
  Race: White | 43 | 13 | 56
  Race: Multiple Races | 2 | 2 | 4
  Race: Unknown | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Main Cohort: THV Dysfunction
Description: Number of patients with THV dysfunction, defined as a non-hierarchical composite of:
  * RVOT/PV Reintervention
  * Moderate or greater total Pulmonic Regurgitation via Transthoracic Echocardiography (TTE)
  * Mean RVOT/PV Gradient >= 35mmHg via TTE
Time Frame: 6 months
Population: Valve implant population, 1 subject did not complete the 6 month follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | TPVR - Main Cohort
Number analyzed (Participants) | 59
Participants | 0

2. Primary Outcome: PDS Registry: Acute PDS Success
Description: Number of patients with acute PDS success, defined as a non-hierarchical composite of:
  * Single THV implanted in the desired location
  * Right ventricle to pulmonary artery (RV-PA) peak-to-peak gradient < 35 mmHg post-THV implantation
  * Less than moderate total pulmonary regurgitation by discharge TTE (or earliest evaluable TTE)
  * Free of SAPIEN 3 / Alterra explant at 24 hours post-implantation
Time Frame: 24 hours
Population: Attempted implant population
Measure: Count of Participants; unit: Participants
Arm/Group | TPVR - PDS Registry
Number analyzed (Participants) | 25
Participants | 22

3. Secondary Outcome: Main Cohort: Improvement in Total Pulmonary Regurgitation From Baseline
Description: Number of patients with improvement in total pulmonary regurgitation
Time Frame: 30 days
Population: Valve implant population
Measure: Count of Participants; unit: Participants
Arm/Group | TPVR - Main Cohort
Number analyzed (Participants) | 60
Participants | 60

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | TPVR - Main Cohort | TPVR - PDS Registry
All-Cause Mortality (participants affected / at risk) | 0/61 | 1/25
Serious Adverse Events (participants affected / at risk) | 8/61 | 5/25
Other Adverse Events (participants affected / at risk) | 35/61 | 11/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TPVR - Main Cohort (N=61) | TPVR - PDS Registry (N=25)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial haemorrhage (Cardiac disorders) | 1 (1) | 0 (0)
Tricuspid valve incompetence (Cardiac disorders) | 2 (2) | 2 (2)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 2 (2)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Prosthetic cardiac valve thrombosis (General disorders) | 1 (1) | 0 (0)
Vascular stent thrombosis (General disorders) | 1 (1) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Venous injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Transvalvular pressure gradient increased (Investigations) | 1 (1) | 0 (0)
Device dislocation (Product Issues) | 1 (1) | 0 (0)
Lead dislodgement (Product Issues) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pelvic venous thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TPVR - Main Cohort (N=61) | TPVR - PDS Registry (N=25)
Tricuspid valve incompetence (Cardiac disorders) | 4 | 0
Venricular extrasystoles (Cardiac disorders) | 10 | 4
Ventricular tachycardia (Cardiac disorders) | 15 | 2
Chest discomfort (General disorders) | 6 | 0
Chest pain (General disorders) | 8 | 6
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 6 | 2
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 4 | 0
Device breakage (Product Issues) | 5 | 3
Deep vein thrombosis (Vascular disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-16): https://cdn.clinicaltrials.gov/large-docs/77/NCT03130777/Prot_SAP_000.pdf